CLINICAL TRIAL: NCT00369278
Title: Multi-center, Open-label, Prospective, Randomized, Parallel Group Study Investigating an Intensified Enteric-coated Mycophenolate Sodium (EC-MPS) Dosing Regimen in Comparison to a Standard Dosing Regimen of EC-MPS in Combination With Cyclosporin Microemulsion and Corticosteroids in de Novo Renal Transplant Patients
Brief Title: Intensified vs. Standard Dose Therapy With Mycophenolate Sodium Plus Cyclosporin Microemulsion and Corticosteroid Combination in Patients With de Novo Renal Transplant Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CERL080ADE12
Record Dates: First submitted 2006-08-25; First posted 2006-08-29 (Estimated); Results first posted 2011-01-12 (Estimated); Last update posted 2011-03-29 (Estimated); Status verified 2011-03

CONDITIONS: Renal Transplantation
Keywords: Renal transplantation, mycophenolate
MeSH Terms: interventions — Mycophenolic Acid

ARMS (2):
- Intensified Mycophenolate sodium (Experimental): Enteric-coated mycophenolate sodium was given according to the following dosing regimen: Day 1-14: 2880 mg/day (2 x 1440 mg), then day 15-42: 2160 mg/day (2 x 1080 mg), then day 43-End of study (month 6): 1440 mg/day (2 x 720 mg). Total duration of treatment was 180 days.
  Interventions: Drug: Enteric-coated mycophenolate sodium (EC-MPS)
- Standard Mycophenolate sodium (Active Comparator): Enteric-coated mycophenolate sodium was given according to the following dosing regimen: Day 1 - End of Study(month 6): 1440 mg/day (2 x 720 mg). Total duration of treatment was 6 months.
  Interventions: Drug: Enteric-coated mycophenolate sodium (EC-MPS)

INTERVENTIONS:
Drug: Enteric-coated mycophenolate sodium (EC-MPS) — Tablets for oral administration
  Other Names: myfortic

SUMMARY:
This study will assess the association of an initially intensified dosing regimen of enteric-coated mycophenolate sodium (EC-MPS) during the first 6 weeks post renal transplantation with acute rejections relative to the rapid achievement of an MPA (mycophenolic acid) exposure of ≥ 40 mg*h/L compared to a standard dosing regimen of EC-MPS. Additionally, this study will assess safety and tolerability of the intensified dosing regimen of EC-MPS. This study will be conducted in 2 stages (Stage I and Stage II).

ELIGIBILITY:
Inclusion criteria

1. Recipients of de novo cadaveric, living unrelated or living related kidney transplants
2. Females capable of becoming pregnant must have a negative serum pregnancy test within 7 days prior to or at baseline, and are required to practice an approved method of birth control for the duration of the study and for a period of 6 weeks following discontinuation of study medication, even where there has been a history of infertility.
3. Patients who are willing and able to participate in the study and from whom written informed consent has been obtained.

Exclusion criteria

1. More than one previous renal transplantation
2. Graft loss due to immunological reasons in the first year after transplantation (in case of secondary transplantation)
3. Multi-organ recipients (e.g., kidney and pancreas) or previous transplant with any other organ, different from kidney
4. Patients receiving a kidney from a non-heart beating donor
5. Patients who are recipients of A-B-O incompatible transplants

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2006-06; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Director — Novartis
Locations (1):
- Novartis Investigational Site, Various Cities, Germany

RESULTS

PARTICIPANT FLOW:
Groups:
- Intensified Mycophenolate Sodium: Enteric-coated mycophenolate sodium was given according to the following dosing regimen: Day 1-14: 2880 mg/day (2 x 1440 mg), then day 15-42: 2160 mg/day (2 x 1080 mg), then day 43-End of study (month 6): 1440 mg/day (2 x 720 mg)
- Standard Mycophenolate Sodium: Enteric-coated mycophenolate sodium was given according to the following dosing regimen: Day 1 - End of Study(month 6): 1440 mg/day (2 x 720 mg)
Period: Overall Study
Arm/Group | Intensified Mycophenolate Sodium | Standard Mycophenolate Sodium
Started | 63 | 65
Completed | 39 | 44
Not Completed | 24 | 21
Not completed — Adverse Event | 14 | 11
Not completed — Unsatisfactory therapeutic effect | 4 | 5
Not completed — Protocol Violation | 2 | 1
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Lost to Follow-up | 1 | 0
Not completed — Graft loss | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intensified Mycophenolate Sodium | Standard Mycophenolate Sodium | Total
Number analyzed (Participants) | 63 | 65 | 128
Age Continuous [Mean (Standard Deviation); unit: years] | 52.4 (12.5) | 50.4 (14.6) | 51.4 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 30 | 59
  Male | 34 | 35 | 69

OUTCOME MEASURES:

1. Primary Outcome: Time to First Occurrence of a Mycophenolic Acid (MPA) Plasma Concentration of ≥ 40 mg*h/L
Description: Non-compartmental MPA pharmacokinetic parameters were derived from individual plasma concentration-time profiles using WinNonLin 5.2 software. The areas under the curve were calculated by means of the linear trapezoidal rule.
Time Frame: Assessed on day 3, 10, 21, 42, 56 and 84
Population: Pharmacokinetic profiles were performed only in patients involved in Phase I of the study. The pharmacokinetic population consisted of 42 participants.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Intensified Mycophenolate Sodium | Standard Mycophenolate Sodium
Number analyzed (Participants) | 23 | 19
Days | 7.00 [5.0 to 23.0] | 43.00 [12.0 to 58.0]

2. Primary Outcome: Time to First Occurrence of Any Treatment Failure During the First 6 Months Post-treatment or at Month 6 Post-treatment
Description: Median time to first occurrence of treatment failure was not reached in this study.
Time Frame: 6 months
Reporting Status: Not Posted

3. Secondary Outcome: Number of Participants With Single Treatment Failures
Description: Rates for all individual components of the primary endpoint 'treatment failure' until day 180:
  * Acute rejection diagnosed by biopsy (BPAR)
  * graft loss
  * death
  * loss to follow up
  * discontinuation from study drug due to lack of efficacy or toxicity (adverse events, every adverse event had to be interpreted as toxicity)
  * conversion to another dosing regimen (conversion to tacrolimus, prograf, etc.)
Time Frame: 6 months
Population: Intent-to-treat population
Measure: Number; unit: Participants
Arm/Group | Intensified Mycophenolate Sodium | Standard Mycophenolate Sodium
Number analyzed (Participants) | 63 | 65
Participants
  Biopsy-proven acute rejection | 2 | 11
  Graft loss | 1 | 2
  Death | 0 | 0
  Loss to follow-up | 1 | 0
  Discontinuation due to lack of efficacy / toxicity | 17 | 15
  Conversion of doses | 8 | 10
  Treated rejections | 13 | 24

4. Secondary Outcome: Rates of Events for Treated Acute Rejection, Death, Graft Loss, or Loss to Follow up on Day 28, Day 84, and Day 180
Description: Due to a small number of events, median time to <event> was not reached.
Time Frame: 6 months
Reporting Status: Not Posted

5. Secondary Outcome: Time to "Event" for the Composite Endpoint as Well as All Individual Components of That Endpoint "Treatment Failure" Including Clinical Rejections
Description: Due to a small number of events, median time to <event> was not reached.
Time Frame: 6 months
Reporting Status: Not Posted

6. Secondary Outcome: Renal Function as Measured by Serum Creatinine
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Intensified Mycophenolate Sodium | Standard Mycophenolate Sodium
Number analyzed (Participants) | 63 | 65
mg/dL
  Baseline | 8.0 (2.7) | 7.8 (2.9)
  End of study | 2.2 (1.5) | 2.6 (2.2)

7. Primary Outcome: Number of Participants With Any Treatment Failure
Description: Treatment failures were defined as a composite endpoint of biopsy proven acute rejection (BPAR), graft loss, and death, loss to follow up and discontinuations from study drug treatment due to lack of efficacy or toxicity (at least one condition must be present) during the first 6 months or until final assessment. Any participants who were suspected of having acute rejection episodes had biopsies performed to prove whether a rejection had occurred. Graft loss was considered as the day the patient started dialysis and was not able to subsequently be removed or the day of graft nephrectomy.
Time Frame: 6 months
Measure: Number; unit: Participants
Arm/Group | Intensified Mycophenolate Sodium | Standard Mycophenolate Sodium
Number analyzed (Participants) | 63 | 65
Participants | 19 | 24

8. Secondary Outcome: Renal Function as Measured by Glomerular Filtration Rate (GFR)
Description: The Glomerular Filtration Rate (GFR) was calculated using the following formulas:
  * Cockcroft-Gault formula: calculation using the participant's age, gender, weight, and serum creatinine levels.
  * MDRD formula: calculation using the participant's age, gender, serum creatinine, urea nitrogen, and albumin levels.
Time Frame: 6 months
Population: Intent-to-treat population for whom data was available. End of Study data was imputed using Last Observation Carried Forward (LOCF).
Measure: Mean (Standard Deviation); unit: ml/min
Arm/Group | Intensified Mycophenolate Sodium | Standard Mycophenolate Sodium
Number analyzed (Participants) | 63 | 65
ml/min
  MDRD formula: Baseline [n=44, 56] | 9.0 (3.9) | 9.4 (3.9)
  MDRD formula: End of study [n=61, 64] | 41.1 (17.1) | 40.6 (24.8)
  Cockcroft-Gault formula: Baseline [n=61, 65] | 12.1 (4.8) | 12.0 (5.0)
  Cockcroft-Gault formula: End of study [n=63, 65] | 52.4 (23.9) | 47.9 (27.1)

ADVERSE EVENTS:
Groups:
- Standard Mycophenolate Sodium: Enteric-coated mycophenolate sodium was given according to the following dosing regimen: Day 1 - End of Study (month 6): 1440 mg/day (2 x 720 mg)
Arm/Group | Intensified Mycophenolate Sodium | Standard Mycophenolate Sodium
Serious Adverse Events (participants affected / at risk) | 44/63 | 40/65
Other Adverse Events (participants affected / at risk) | 62/63 | 63/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intensified Mycophenolate Sodium (N=63) | Standard Mycophenolate Sodium (N=65)
Anaemia (Blood and lymphatic system disorders) | 2 | 0
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 1
Tricuspid valve incompetence (Cardiac disorders) | 0 | 1
Wolff-Parkinson-White syndrome (Cardiac disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 4 | 1
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1
Duodenitis (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 2
Inguinal hernia (Gastrointestinal disorders) | 0 | 1
Inguinal hernia, obstructive (Gastrointestinal disorders) | 0 | 1
Intra-abdominal haematoma (Gastrointestinal disorders) | 1 | 0
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 1 | 0
Large intestine perforation (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1
Reflux oesophagitis (Gastrointestinal disorders) | 0 | 1
Small intestinal perforation (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1
Catheter related complication (General disorders) | 0 | 1
Impaired healing (General disorders) | 1 | 0
Multi-organ failure (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Transplant rejection (Immune system disorders) | 0 | 2
Abdominal abscess (Infections and infestations) | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 1
Cytomegalovirus gastritis (Infections and infestations) | 1 | 0
Cytomegalovirus infection (Infections and infestations) | 2 | 1
Enterococcal infection (Infections and infestations) | 1 | 1
Escherichia bacteraemia (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Gastroenteritis clostridial (Infections and infestations) | 1 | 0
Gastroenteritis norovirus (Infections and infestations) | 2 | 1
Gastrointestinal infection (Infections and infestations) | 0 | 1
Haematoma infection (Infections and infestations) | 1 | 0
Human polyomavirus infection (Infections and infestations) | 1 | 1
Infected lymphocele (Infections and infestations) | 0 | 2
Infection (Infections and infestations) | 2 | 1
Oesophageal candidiasis (Infections and infestations) | 0 | 1
Otitis media (Infections and infestations) | 1 | 0
Perinephric abscess (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 4 | 0
Renal abscess (Infections and infestations) | 0 | 1
Renal cyst infection (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Staphylococcal infection (Infections and infestations) | 1 | 0
Tracheobronchitis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 5 | 9
Urosepsis (Infections and infestations) | 1 | 4
Wound abscess (Infections and infestations) | 1 | 0
Wound infection (Infections and infestations) | 2 | 0
Wound infection bacterial (Infections and infestations) | 1 | 0
Wound infection staphylococcal (Infections and infestations) | 1 | 0
Anastomotic leak (Injury, poisoning and procedural complications) | 1 | 0
Arteriovenous graft thrombosis (Injury, poisoning and procedural complications) | 2 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 1
Complications of transplanted kidney (Injury, poisoning and procedural complications) | 2 | 3
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1
Graft loss (Injury, poisoning and procedural complications) | 2 | 2
Incisional hernia (Injury, poisoning and procedural complications) | 1 | 1
Perirenal haematoma (Injury, poisoning and procedural complications) | 0 | 2
Post procedural urine leak (Injury, poisoning and procedural complications) | 2 | 1
Seroma (Injury, poisoning and procedural complications) | 0 | 1
Shunt aneurysm (Injury, poisoning and procedural complications) | 1 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Transplant failure (Injury, poisoning and procedural complications) | 0 | 5
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 1
Blood creatinine increased (Investigations) | 9 | 6
Haemoglobin decreased (Investigations) | 0 | 1
Calciphylaxis (Metabolism and nutrition disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hypervolaemia (Metabolism and nutrition disorders) | 0 | 1
Cerebral infarction (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Migraine (Nervous system disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 1
Uraemic encephalopathy (Nervous system disorders) | 0 | 1
Delirium (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 1 | 0
Hallucination, visual (Psychiatric disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 1
Renal artery occlusion (Renal and urinary disorders) | 1 | 0
Renal artery stenosis (Renal and urinary disorders) | 2 | 0
Renal failure (Renal and urinary disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 4 | 5
Ureteral necrosis (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 2 | 1
Urinary tract obstruction (Renal and urinary disorders) | 1 | 1
Urinoma (Renal and urinary disorders) | 1 | 2
Vesicoureteric reflux (Renal and urinary disorders) | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1
Pelvic congestion (Reproductive system and breast disorders) | 2 | 2
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Skin inflammation (Skin and subcutaneous tissue disorders) | 1 | 0
Pneumatic compression therapy (Surgical and medical procedures) | 0 | 1
Wound treatment (Surgical and medical procedures) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 2
Femoral arterial stenosis (Vascular disorders) | 1 | 0
Haematoma (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 2 | 1
Lymphocele (Vascular disorders) | 4 | 3
Peripheral artery aneurysm (Vascular disorders) | 1 | 0
Peripheral artery dissection (Vascular disorders) | 1 | 0
Shock (Vascular disorders) | 0 | 1
Shock haemorrhagic (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Intensified Mycophenolate Sodium (N=63) | Standard Mycophenolate Sodium (N=65)
Anaemia (Blood and lymphatic system disorders) | 16 | 19
Leukopenia (Blood and lymphatic system disorders) | 12 | 14
Thrombocytopenia (Blood and lymphatic system disorders) | 4 | 1
Abdominal pain (Gastrointestinal disorders) | 11 | 5
Constipation (Gastrointestinal disorders) | 19 | 15
Diarrhoea (Gastrointestinal disorders) | 19 | 23
Dyspepsia (Gastrointestinal disorders) | 4 | 0
Flatulence (Gastrointestinal disorders) | 13 | 7
Nausea (Gastrointestinal disorders) | 23 | 19
Vomiting (Gastrointestinal disorders) | 16 | 16
Oedema (General disorders) | 16 | 14
Oedema peripheral (General disorders) | 15 | 16
Pain (General disorders) | 1 | 4
Pyrexia (General disorders) | 3 | 8
BK virus infection (Infections and infestations) | 4 | 1
Cytomegalovirus infection (Infections and infestations) | 2 | 7
Nasopharyngitis (Infections and infestations) | 3 | 8
Pneumonia (Infections and infestations) | 1 | 7
Rhinitis (Infections and infestations) | 4 | 5
Urinary tract infection (Infections and infestations) | 24 | 26
Complications of transplanted kidney (Injury, poisoning and procedural complications) | 20 | 22
Procedural pain (Injury, poisoning and procedural complications) | 3 | 4
Wound complication (Injury, poisoning and procedural complications) | 9 | 13
Wound dehiscence (Injury, poisoning and procedural complications) | 7 | 9
Blood creatinine increased (Investigations) | 7 | 12
Blood glucose increased (Investigations) | 5 | 2
C-reactive protein increased (Investigations) | 7 | 1
Haemoglobin decreased (Investigations) | 4 | 1
Weight increased (Investigations) | 4 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 5 | 6
Hypercholesterolaemia (Metabolism and nutrition disorders) | 7 | 6
Hyperkalaemia (Metabolism and nutrition disorders) | 9 | 9
Hyperphosphataemia (Metabolism and nutrition disorders) | 4 | 6
Hyperuricaemia (Metabolism and nutrition disorders) | 4 | 5
Hypocalcaemia (Metabolism and nutrition disorders) | 19 | 14
Hypokalaemia (Metabolism and nutrition disorders) | 23 | 31
Hypomagnesaemia (Metabolism and nutrition disorders) | 6 | 5
Hypophosphataemia (Metabolism and nutrition disorders) | 13 | 10
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 5
Muscle spasms (Musculoskeletal and connective tissue disorders) | 7 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 5
Headache (Nervous system disorders) | 8 | 9
Tremor (Nervous system disorders) | 4 | 3
Sleep disorder (Psychiatric disorders) | 11 | 12
Bladder pain (Renal and urinary disorders) | 6 | 9
Dysuria (Renal and urinary disorders) | 6 | 3
Haematuria (Renal and urinary disorders) | 7 | 5
Residual urine (Renal and urinary disorders) | 4 | 1
Urinary retention (Renal and urinary disorders) | 6 | 2
Urinary tract obstruction (Renal and urinary disorders) | 1 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 7
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 8
Haematoma (Vascular disorders) | 0 | 5
Hypertension (Vascular disorders) | 10 | 4
Hypotension (Vascular disorders) | 8 | 3
Lymphocele (Vascular disorders) | 4 | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.